CLINICAL TRIAL: NCT00739739
Title: A Phase 2, 12 Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Proof Of Concept Study Evaluating The Efficacy And Safety Of PD 0299685 For The Treatment Of Symptoms Associated With Interstitial Cystitis/Painful Bladder Syndrome.
Brief Title: An Effectiveness And Safety Study Of PD 0299685 For The Treatment Of Symptoms Associated With Interstitial Cystitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4291043
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PD 0299685 15mg (Experimental)
  Interventions: Drug: PD 0299685 at 15mg BID
- PD 0299685 30mg (Experimental)
  Interventions: Drug: PD 0299685 at 30mg BID
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo for PD 0299685

INTERVENTIONS:
Drug: PD 0299685 at 15mg BID — 5 mg Capsules, 3 to be taken in the morning and at bedtime for the duration of the study
  Arms: PD 0299685 15mg
Drug: PD 0299685 at 30mg BID — 10mg Capsules, 3 to be taken in the morning and at bedtime for the duration of the study. Initial 2 week titration period at 15mg BID.
  Arms: PD 0299685 30mg
Drug: placebo for PD 0299685 — Capsules identical in appearance to PD 0299685, 3 to be taken in the morning and at bedtime for the duration of the study
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether PD 0299685 is effective in the treatment of symptoms associated with interstitial cystitis/painful bladder syndrome, such as pain, urinary urgency and frequency. At the same time assess the drug's safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age with moderate to severe interstitial cystitis defined by pain score.
* Women must not be pregnant or lactating, They may be post-menopausal, surgically sterilized or using an appropriate method of contraception.

Exclusion Criteria:

* History of interstitial cystitis less than 6 months
* History of current or recurrent urinary tract infections, or genitourinary cancer
* Any previous urinary diversion procedure with or without bladder removal, bladder augmentation
* Use of certain drugs given into the bladder up to 1 month prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) score. | 12 WEEKS
Change from baseline in worst daily pain severity score as measured by an 11-point Numerical Rating Scale (NRS). | 12 WEEKS

SECONDARY OUTCOMES:
Micturition Diary Variables including frequency, urgency, nocturnal frequency, incontinence episodes. | 12 weeks
ICSI at other time points | 12 weeks
Interstitial Cystitis Problem Index (ICPI) | 12 weeks
Pelvic pain Urgency Frequency score (PUF) | 12 weeks
Epworth Sleepiness Scale (ESS) | 12 Weeks
Columbia-Suicide Severity Rating Scale (C-SSRS) | 15 Weeks
Adverse events | 15 Weeks
Physical examination | 14 Weeks
Vital signs and weight | 15 Weeks
ECG | 14 Weeks
Residual urine volume measurement | 14 Weeks
Global Response assessment (GRA) | 12 Weeks
Patient Reported Treatment Impact (PRTI) | 12 Weeks
Treatment failures | 12 Weeks
Average and worst daily pain score at other time points as measured by an 11-point NRS. | 12 Weeks
Sleep disturbance and sexual activity pain. | 12 Weeks
Clinical laboratory tests | 14 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- United States (23):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Goodyear, Arizona
  - Pfizer Investigational Site, Litchfield Park, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Glendora, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Brighton, Massachusetts
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Garden City, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Burlington, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, West Chester, Ohio
  - Pfizer Investigational Site, Bethany, Oklahoma
  - Pfizer Investigational Site, State College, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Spokane, Washington
- Canada (6):
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Pfizer Investigational Site, Herlev, Denmark
- Finland (5):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Kouvola
  - Pfizer Investigational Site, OYS
  - Pfizer Investigational Site, Seinäjoki
  - Pfizer Investigational Site, Tampere
- France (6):
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Nîmes
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Strasbourg
- Germany (2):
  - Pfizer Investigational Site, Homburg
  - Pfizer Investigational Site, München

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597
- [Derived] Nickel JC, Crossland A, Davis E, Haab F, Mills IW, Rovner E, Scholfield D, Crook T. Investigation of a Ca2+ channel alpha2delta ligand for the treatment of interstitial cystitis: results of a randomized, double-blind, placebo controlled phase II trial. J Urol. 2012 Sep;188(3):817-23. doi: 10.1016/j.juro.2012.05.010. Epub 2012 Jul 19. PMID 22818144